CLINICAL TRIAL: NCT05922839
Title: Zanubrutinib in Relapsed or Refractory Warm Autoimmune Hemolytic Anemia: a Prospective Cohort Study
Brief Title: Zanubrutinib in the Treatment of Relapsed/Refractory wAIHA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chen Miao (Other)
Responsible Party: Sponsor-Investigator, Chen Miao, associate professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zanubrutinib-1
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Warm Autoimmune Hemolytic Anemia
Keywords: warm autoimmune hemolytic anemia; Zanubrutinib
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib in the Treatment of Relapsed/Refractory wAIHA (Experimental): Zanubrutinib 160mg, orally, twice daily, for a minimum of 3 months For effective patients, continue to use for 2 years after achieving optimal therapeutic effect.
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib 160mg, orally, twice daily, for a minimum of 3 months, and for effective patients, continue to use for 2 years after achieving optimal therapeutic effect.

SUMMARY:
Autoimmune hemolytic anemia (AIHA) is a rare and heterogeneous disorder characterized by the destruction of red blood cells through warm or cold antibodies. Glucocorticoid (combined with rituximab) is the first-line treatment.

However, the recurrence rate is very high and some patients may not respond to steroids. Second-line therapies include cyclosporine A (CsA), cyclophosphamide, rituximab, azathioprine, and even splenectomy.

Bruton's tyrosine kinase (BTK) plays a crucial role in the signaling pathway of B-cell receptor (BCR), and has been found to be a major source of pathogenic signal transduction for various lymphoproliferative malignancies. The activity of BTK is related to the occurrence and progression of various B-cell lymphomas. Currently, BTK inhibitors are widely used in the treatment of B-cell lymphomas, including chronic lymphocytic leukemia (CLL), mantle cell lymphoma (MCL), Waldenstrom's macroglobulinemia (WM), and other B-cell lymphomas, showing significant efficacy. BTK affects the production of messenger molecules and regulates the BCR signaling pathway, causing B cells to transform into self-reactive B cells, which can trigger autoimmune diseases. Current research has shown that BTK activity increases in several autoimmune diseases, including systemic lupus erythematosus (SLE) and rheumatoid arthritis (RA) . Therefore, BTK inhibitors (BTKi) are important for the treatment of autoimmune diseases.

Ibrutinib, one kind of BTKi, has been proven to treat secondary autoimmune hemolytic anemia (AIHA) in CLL and control CLL progression, and is an effective drug for treating lymphoma-associated AIHA . One kind of second-generation selective BTKi, acalabrutinib, can also reduce the incidence of AIHA in relapsed or refractory CLL patients. Currently, phase-II clinical studies exploring the treatment of AIHA using Ibrutinib, acalabrutinib, and rilzabrutinib, another BTKi, are underway.

Zanubrutinib (BGB-3111, Brukinsa®, BeiGene) is a second-generation irreversible BTKi developed by Chinese company BeiGene. Compared to Ibrutinib, zanubrutinib has shown stronger effective activity and higher selectivity towards BTK, and weaker effects on other targets such as TEC, EGFR, and Src families, with low off-target side effects. Its efficacy, durability, oral absorption, and targeting are better than those of Ibrutinib. Zanubrutinib is approved for the treatment of various B-cell lymphomas, and clinical trials have shown excellent efficacy and tolerability in CLL and WM patients. In previously treated CLL patients, zanubrutinib exhibits better efficacy and safety than Ibrutinib. Currently, phase II clinical studies of zanubrutinib in ITP, antiphospholipid syndrome, IgG4-related immune diseases, and active proliferative lupus nephritis are underway. The therapeutic effect of zanubrutinib on refractory warm autoimmune hemolytic anemia, is worth exploring through exploratory research.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Confirmed diagnosis of wAIHA or Evans syndrome, primary or secondary to connective tissue disease. If it is secondary, there are no other treatment indications for systemic involvement of primary connective tissue disease.
3. No response or relapse after glucocorticoid treatment.
4. Baseline liver and kidney function (ALT, AST, Cr) is less than 2 times the normal range.
5. Consent to sign the informed consent form.

Exclusion Criteria:

1. Other important organ involvement in connective tissue disease.
2. Uncontrolled infection or bleeding with standard treatment.
3. Active HIV, HCV or HBV infection uncontrolled with standard treatment.
4. Concurrent uncontrolled advanced malignant tumors or lymphoma.
5. The subject is receiving any of the following drugs and has not met the following conditions of stable drug treatment duration at a fixed dose during screening: corticosteroids for at least 4 weeks; iron, vitamin B12 or folic acid for at least 4 weeks;
6. Liver cirrhosis or portal hypertension.
7. Pregnant or lactating women.
8. Participation in other clinical trials within the last 3 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 3/6 months
  ORR defined as the proportion of patients who met the criteria of either complete response (CR) or partial response (PR)
Complete response rate (CRR) | 3/6 months
  CRR defined as the proportion of patients who met the criteria of complete response.

SECONDARY OUTCOMES:
Relapse rate | 3/6 months
  Relapse rate defined as the proportion of patients whose response shift from PR or CR to no response (NR).
Adverse events | 3/6 months
  Safety analyses include assessments of the incidence and severity of adverse events; all adverse events that occurred or worsened during the treatment period will be reported, as well as adverse events that occurred later but are considered by the investigator to be related to the trial drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jager U, Barcellini W, Broome CM, Gertz MA, Hill A, Hill QA, Jilma B, Kuter DJ, Michel M, Montillo M, Roth A, Zeerleder SS, Berentsen S. Diagnosis and treatment of autoimmune hemolytic anemia in adults: Recommendations from the First International Consensus Meeting. Blood Rev. 2020 May;41:100648. doi: 10.1016/j.blre.2019.100648. Epub 2019 Dec 5. PMID 31839434
- [Background] Birgens H, Frederiksen H, Hasselbalch HC, Rasmussen IH, Nielsen OJ, Kjeldsen L, Larsen H, Mourits-Andersen T, Plesner T, Ronnov-Jessen D, Vestergaard H, Klausen TW, Schollkopf C. A phase III randomized trial comparing glucocorticoid monotherapy versus glucocorticoid and rituximab in patients with autoimmune haemolytic anaemia. Br J Haematol. 2013 Nov;163(3):393-9. doi: 10.1111/bjh.12541. Epub 2013 Aug 24. PMID 23981017
- [Background] Zarrin AA, Bao K, Lupardus P, Vucic D. Kinase inhibition in autoimmunity and inflammation. Nat Rev Drug Discov. 2021 Jan;20(1):39-63. doi: 10.1038/s41573-020-0082-8. Epub 2020 Oct 19. PMID 33077936
- [Background] Ringheim GE, Wampole M, Oberoi K. Bruton's Tyrosine Kinase (BTK) Inhibitors and Autoimmune Diseases: Making Sense of BTK Inhibitor Specificity Profiles and Recent Clinical Trial Successes and Failures. Front Immunol. 2021 Nov 3;12:662223. doi: 10.3389/fimmu.2021.662223. eCollection 2021. PMID 34803999
- [Background] McDonald C, Xanthopoulos C, Kostareli E. The role of Bruton's tyrosine kinase in the immune system and disease. Immunology. 2021 Dec;164(4):722-736. doi: 10.1111/imm.13416. Epub 2021 Oct 4. PMID 34534359
- [Background] Liubchenko GA, Appleberry HC, Striebich CC, Franklin KE, Derber LA, Holers VM, Lyubchenko T. Rheumatoid arthritis is associated with signaling alterations in naturally occurring autoreactive B-lymphocytes. J Autoimmun. 2013 Feb;40:111-21. doi: 10.1016/j.jaut.2012.09.001. Epub 2012 Oct 8. PMID 23058039
- [Background] Iwata S, Tanaka Y. B-cell subsets, signaling and their roles in secretion of autoantibodies. Lupus. 2016 Jul;25(8):850-6. doi: 10.1177/0961203316643172. PMID 27252261
- [Background] Montillo M, O'Brien S, Tedeschi A, Byrd JC, Dearden C, Gill D, Brown JR, Barrientos JC, Mulligan SP, Furman RR, Cymbalista F, Plascencia C, Chang S, Hsu E, James DF, Hillmen P. Ibrutinib in previously treated chronic lymphocytic leukemia patients with autoimmune cytopenias in the RESONATE study. Blood Cancer J. 2017 Feb 3;7(2):e524. doi: 10.1038/bcj.2017.5. No abstract available. PMID 28157216
- [Background] Rogers KA, Ruppert AS, Bingman A, Andritsos LA, Awan FT, Blum KA, Flynn JM, Jaglowski SM, Lozanski G, Maddocks KJ, Byrd JC, Woyach JA, Jones JA. Incidence and description of autoimmune cytopenias during treatment with ibrutinib for chronic lymphocytic leukemia. Leukemia. 2016 Feb;30(2):346-50. doi: 10.1038/leu.2015.273. Epub 2015 Oct 7. PMID 26442611
- [Background] Manda S, Dunbar N, Marx-Wood CR, Danilov AV. Ibrutinib is an effective treatment of autoimmune haemolytic anaemia in chronic lymphocytic leukaemia. Br J Haematol. 2015 Sep;170(5):734-6. doi: 10.1111/bjh.13328. Epub 2015 Feb 25. No abstract available. PMID 25716177
- [Background] Galinier A, Delwail V, Puyade M. Ibrutinib Is Effective in the Treatment of Autoimmune Haemolytic Anaemia in Mantle Cell Lymphoma. Case Rep Oncol. 2017 Jan 27;10(1):127-129. doi: 10.1159/000456002. eCollection 2017 Jan-Apr. PMID 28203175
- [Background] Byrd JC, Wierda WG, Schuh A, Devereux S, Chaves JM, Brown JR, Hillmen P, Martin P, Awan FT, Stephens DM, Ghia P, Barrientos J, Pagel JM, Woyach JA, Burke K, Covey T, Gulrajani M, Hamdy A, Izumi R, Frigault MM, Patel P, Rothbaum W, Wang MH, O'Brien S, Furman RR. Acalabrutinib monotherapy in patients with relapsed/refractory chronic lymphocytic leukemia: updated phase 2 results. Blood. 2020 Apr 9;135(15):1204-1213. doi: 10.1182/blood.2018884940. PMID 31876911
- [Background] Robak E, Robak T. Bruton's Kinase Inhibitors for the Treatment of Immunological Diseases: Current Status and Perspectives. J Clin Med. 2022 May 16;11(10):2807. doi: 10.3390/jcm11102807. PMID 35628931
- [Background] Guo Y, Liu Y, Hu N, Yu D, Zhou C, Shi G, Zhang B, Wei M, Liu J, Luo L, Tang Z, Song H, Guo Y, Liu X, Su D, Zhang S, Song X, Zhou X, Hong Y, Chen S, Cheng Z, Young S, Wei Q, Wang H, Wang Q, Lv L, Wang F, Xu H, Sun H, Xing H, Li N, Zhang W, Wang Z, Liu G, Sun Z, Zhou D, Li W, Liu L, Wang L, Wang Z. Discovery of Zanubrutinib (BGB-3111), a Novel, Potent, and Selective Covalent Inhibitor of Bruton's Tyrosine Kinase. J Med Chem. 2019 Sep 12;62(17):7923-7940. doi: 10.1021/acs.jmedchem.9b00687. Epub 2019 Aug 19. PMID 31381333